CLINICAL TRIAL: NCT06967649
Title: Prospective Longitudinal Clinical Study for the Evaluation of Peri-implant Tissue and Osseointegration After Rehabilitation With Osseointegrated Implants
Acronym: Dental Implant
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Priscila Ladeira Casado, PhD in Morphology , Professor and Researcher at the Universidade Federal Fluminense, Universidade Federal Fluminense
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DENTAL IMPLANTS EVALUATION
Record Dates: First submitted 2025-05-03; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Osseointegration Failure of Dental Implant; Periimplantitis; Peri-Implant Tissues; Peri-Implant Health; Peri-implant Soft Tissue Healing; Implant Survival Using Immediate Loading Protocol; Dental Implant Stability; Prospective Study; Osseointegration
Keywords: PERI-IMPLANT HEALTH; Dental implant survival rate; DENTAL IMPLANT; prospective study; osseointegration
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMPLANT PLACEMENT (Active Comparator): Research participants will undergo clinical and prosthetic planning (reverse planning), including clinical-tomographic examinations and complementary tests, such as biochemical blood analysis and, when necessary, surgical risk assessment, according to the UFF Implant Dentistry specialization course protocol. The surgical technique, type of implant installed, and selected prosthetic components will follow the manufacturer's recommendations (SIN Implant System, São Paulo, Brazil), always considering treatment options for optimal patient rehabilitation.
  Interventions: Device: TITANIUM IMPLANT

INTERVENTIONS:
Device: TITANIUM IMPLANT — The surgical technique, type of implant installed, and selected prosthetic components will follow the manufacturer's recommendations (SIN Implant System, São Paulo, Brazil), always considering treatment options for optimal patient rehabilitation.

SUMMARY:
The success of rehabilitation with osseointegrated implants is associated with numerous factors, including patient characteristics, installed implants, proper planning, and the prosthetic connections used. In the long term, success is closely related to the clinical radiographic follow-up of the implanted region and the identification of intrinsic or extrinsic factors that may interfere with implant survival. Therefore, the objective of this study is to evaluate, through clinical and radiographic analysis, the peri-implant tissues and prosthetic connections of research participants rehabilitated with osseointegrated implants at the Implant Dentistry Clinic of the Federal Fluminense University, over a period of 5 years. This will be a double-blind longitudinal study. A total of 148 research participants will be selected, respecting the inclusion criteria: completion of surgical-prosthetic planning by the Implant Dentistry Clinic team at UFF, including osseointegrated implants and prosthetic components manufactured by SIN Implant System (São Paulo, Brazil); agreeing to and signing the informed consent form, being willing to be monitored for a period of 5 years; systemically healthy patients who do not use antiresorptive and antiangiogenic drugs; patients with a plaque index <20% (Ainamo & Bay 1975) and bleeding on probing <20% (Muhlemann & Son 1971) at the start of the study. Participants will undergo clinical and radiographic analysis of peri-implant tissues and prosthetic connections at the following intervals: up to 7 days after implant installation (Time 0), at the time of prosthesis installation (Time 1), 6 months after prosthesis installation (Time 2), and 1 to 5 years after prosthesis installation (Times 3, 4, 5, 6, and 7, respectively). It is expected that this longitudinal study will lead to a better understanding of the factors influencing peri-implant bone loss and long-term success.

DETAILED DESCRIPTION:
Selection of Research Participants Patients treated in the Implant Dentistry specialization course at FO-UFF, who undergo implant dentistry planning and receive rehabilitative treatment with endosseous implants, will be invited to participate in the research, provided they meet the inclusion criteria.

* Inclusion Criteria: Completion of surgical-prosthetic planning by the Implant Dentistry Clinic team at UFF, including osseointegrated implants and prosthetic components manufactured by SIN Implant System (São Paulo, Brazil); agreement to sign the informed consent form and willingness to be monitored for a period of 5 years, following the previously established course clinic protocol; systemically healthy patients who do not use antiresorptive and antiangiogenic drugs; patients with a plaque index <20% (Ainamo & Bay 1975) and bleeding on probing <20% (Muhlemann & Son 1971) at the start of the study.
* Exclusion Criteria: Patients undergoing rehabilitation with implants from different systems and/or not performed at the UFF Implant Dentistry specialization clinic; patients unable to attend radiographic follow-up over 5 years; patients unable to respond to questions in clinical analysis and satisfaction survey forms; presence of systemic conditions preventing the surgical procedure for dental implant installation; presence of metabolic bone disorders; presence of untreated or uncontrolled chronic or aggressive periodontitis; pregnant or lactating women.

Based on these criteria, a total of 148 research participants will be included and followed for 72 months (6 years).

Installation of Osseointegrated Implants Research participants will undergo clinical and prosthetic planning (reverse planning), including clinical-tomographic examinations and complementary tests, such as biochemical blood analysis and, when necessary, surgical risk assessment, according to the UFF Implant Dentistry specialization course protocol. The surgical technique, type of implant installed, and selected prosthetic components will follow the manufacturer's recommendations (SIN Implant System, São Paulo, Brazil), always considering treatment options for optimal patient rehabilitation.

1.1. Clinical Evaluation The clinical evaluation will include detailed anamnesis, assessment of participant satisfaction, peri-implant clinical examination, and evaluation of prosthetic connections over 5 years (Appendix 2). Clinical data will be updated throughout the study evaluations (Table 1) to analyze possible changes in satisfaction or peri-implant tissue condition.

Immediately after implant installation, primary stability will be assessed, with implants considered stable if inserted with a torque above 30 N/cm, without any mobility (Atsumi et al., 2007).

The peri-implant clinical examination will be performed on the mesial, distal, buccal, and lingual surfaces of each implant using a North Carolina periodontal probe (PCPUNC15-6) Hufriedy do Brasil. The following clinical parameters will be observed: spontaneous bleeding, mobility presence; plaque and calculus presence; keratinized tissue presence; peri-implant biotype; mucosal color changes; presence of swollen areas; implant thread exposure; percussion sensitivity; implant function duration; peri-implant probing depth; bleeding on probing and/or suppuration after gentle probing; percussion sound; bone loss presence beyond what is observed after bone remodeling, as well as anamnesis for health data collection (Appendix 2).

Implants will be considered successful if they have no clinical mobility, absence of clinical symptoms such as swelling, paresthesia, or pain, no damage to surrounding structures, no damage to implant or components, no peri-implant radiolucency, and minimal crest bone height loss, according to Albrektsson et al. (1994) and Misch et al. (2008).

1.2. Radiographic Evaluation The radiographic examination consists of digital periapical radiography using the Shick Elite Digital Indicator Cone radiographic positioner - Indusbello. The choice of this radiographic technique is based on literature data highlighting its advantages, such as reduced magnification and distortion, better resolution, and image detail. All radiographic images will be taken using the same X-ray machine by a single operator, different from the operator conducting the clinical analyses. During the radiographic imaging, participants will wear a lead apron and thyroid collar, in compliance with Federal Ordinance 453/98 (01/06/1998).

The radiographic examination will be performed on all research participants, along with clinical exams at the intervals described in Table 1.

Examiner Calibration:

For the radiographic evaluations, a dentist will be calibrated to measure the distance from the implant platform to the first point of contact between bone and implant on the mesial and distal surfaces, using tools such as zoom and digital measurement in a specific image software (ImageProPlus® - Media Cybernetics, Inc.401 N. Washington Street, Suite 350 - Rockville, MD 20850 - United States). After 24 hours, the measurements will be repeated to verify the consistency of results and obtain calibration correlation.

The radiographs will be digitized and evaluated using the image software (ImageProPlus®) for the following parameter: Height of the Marginal Peri-implant Bone Crest: linear measurement of the distance from the implant platform to the first point of contact between bone and implant on the mesial and distal surfaces.

Physiological bone loss will be characterized by considering normal bone loss of one millimeter during the first year after implant placement and 0.2 mm per subsequent year, in accordance with the osseointegration period. Thus, the total amount of bone loss will be calculated based on diagnostic radiography, compared to the clinical implant placement protocol. If total bone loss exceeds 1 mm and 0.2 mm per year, the region will be diagnosed with peri-implantitis (Roos et al., 1997).

1.3. Tomographic Evaluation The tomographic examination will be conducted in partnership with a radiology clinic to be defined, using cone beam computed tomography (CBCT).

According to Monje et al. 2019, measurement accuracy is influenced by defect size and image quality. Intraoral radiography provides a two-dimensional image of the peri-implant bone, describing mesial and distal bone sites; however, it may underestimate incipient lesions and intraosseous defects. Geometric distortions and anatomical overlaps may also occur. In cases where three-dimensional bone visualization is necessary, CBCT can be the alternative.

Participants diagnosed with pathological bone loss radiographically will undergo a tomographic examination at the peri-implant diseased site, aiming to obtain a three-dimensional anatomical image of the bone with its peri-implant defect, serving as a comparison and analysis for the treatment option to be offered.

1.4. Statistical Analysis Prisma GraphPad 6.0 software (GraphPad Software, La Jolla, CA, USA) will be used for all statistical analyses. The distribution type of numerical variables, including clinical data and radiographic measurements, will be assessed using the Shapiro-Wilk test. Student's t-tests or Mann-Whitney tests will be applied for normally or non-normally distributed data, respectively. Paired analyses will be conducted for characteristic comparisons with a significance level of 0.05% (p<0.05). Logistic regression will evaluate the correlation of analyzed factors over the years and the success of rehabilitation.

ELIGIBILITY:
Inclusion Criteria: Completion of surgical-prosthetic planning by the Implant Dentistry Clinic team at UFF, including osseointegrated implants and prosthetic components manufactured by SIN Implant System (São Paulo, Brazil); agreement to sign the informed consent form and willingness to be monitored for a period of 5 years, following the previously established course clinic protocol; systemically healthy patients who do not use antiresorptive and antiangiogenic drugs; patients with a plaque index <20% (Ainamo & Bay 1975) and bleeding on probing <20% (Muhlemann & Son 1971) at the start of the study.

-

Exclusion Criteria: Patients undergoing rehabilitation with implants from different systems and/or not performed at the UFF Implant Dentistry specialization clinic; patients unable to attend radiographic follow-up over 5 years; patients unable to respond to questions in clinical analysis and satisfaction survey forms; presence of systemic conditions preventing the surgical procedure for dental implant installation; presence of metabolic bone disorders; presence of untreated or uncontrolled chronic or aggressive periodontitis; pregnant or lactating women.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
PRIMARY IMPLANT STABILITY | From enrollment to the end of treatment at 6 months
  Data on the clinical and radiographic characteristics of the different installed implants and the short-term stability of their prosthetic connections will be obtained. Over the years of evaluation, there may be better recognition of the factors influencing peri-implant bone loss and long-term success.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal Fluminense, Niterói, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No